CLINICAL TRIAL: NCT04677231
Title: Evaluation of Long-term Health Status and Quality of Life in Adult Survivors With Philadelphia-negative Acute Lymphoblastic Leukemia/Lymphoma Treated With an Intensive Pediatric or Pediatric-inspired Protocol
Acronym: EQUAALL01
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P150969J
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall survival of adult patients (15-59y) with Philadelphia-negative acute lymphoblastic leukemia/lymphoma (ALL/LL) was dramatically improved by the use of full pediatric or pediatric-inspired protocols (GRAALL2003/05-LL03-FRALLE2000) that aimed to reduce the risk of relapse by adopting more intensive chemotherapeutical schedule. This approach led to a global improvement in overall survival (5y-OS, 57%) whatever patient age but was responsible for an excess of treatment-related mortality in patients older than 45 years (5y-TRM in patients > 45y, 19%). Pediatric longitudinal studies pointed out that long term leukemia survivors have an increased risk of developing specific adverse events like dysmetabolic syndrome, obesity, decreased fertility, organ dysfunction, osseous events, or impaired cognitive functions. This study aims to evaluate the impact in term of long-term events and QoL in adult patients that received an intensified therapeutic approach recently implemented in adult cooperative groups. The main objective of this study is to evaluate the prevalence of late effects in adult patients treated 10 years ago for ALL/LL with an intensified pediatric-inspired protocol (GRAALL2003/05-LL03-FRALLE2000) that exposed patients to increased cumulative doses of chemotherapy, central nervous system irradiation or w/o allogeneic transplant after total body irradiation-based regimen w/o boost irradiation on central nevous system. One of the secondary endpoint of the study is to assess quality of life of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Philadelphia-negative ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
* Patients older than 15 years old and less than 60 years old at diagnosis
* Patient with a follow-up from first complete remission of more than 10 years,
* Patient who gave informed signed consent for baseline examination

Exclusion Criteria:

* Patient who experienced ALL/LL relapse within the 5 past years.
* Philadelphia positive ALL patients

Ages: 25 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 15-59y at diagnosis treated ten years ago for a Ph1-negative acute lymphoblastic leukemia/lymphoma (ALL/LL)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of adverse events | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
  This is a binary, composite, endpoint, including any of the following adverse events:
  * metabolic troubles (dysmetabolic syndrome, dyslipidemia, diabetes)
  * osseous events /osteoporosis
  * cardiac and vascular troubles
  * neurologic troubles
  * lung dysfunctions
  * endocrinal troubles

SECONDARY OUTCOMES:
Prevalence of metabolic troubles | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
  Metabolic troubles will be defined as dysmetabolic syndrome or dyslipidemia or diabetes
Prevalence of osseous events | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
Prevalence of cardiac and vascular troubles | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
Prevalence of neurologic troubles | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
Prevalence of lung dysfunctions | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
Prevalence of endocrinal troubles | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
Quality of Life | Up to 3 months post inclusion (10 years from first complete remission of a ALL or LL treated in or according to a pediatric-like or pediatric-inspired protocol (GRAALL03/05-LL03-FRALLE2000) with or without allogeneic transplant.
  Quality of life will be assess using the SF36-questionnaire. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are grouped into three categories: functional status, well-being, overall health assessment. In two dimensions, the answer is binary (yes / no) and in the other 6 in ordinal quality (3 to 6 possible answers). For each dimension, the scores for the different items are coded and then summed and transformed linearly on a scale ranging from 0 to 100. A physical composite score and a mental composite score can be calculated according to an established algorithm

IPD SHARING:
Plan to Share IPD: Undecided